CLINICAL TRIAL: NCT00473291
Title: Vibration Response Imaging (VRI) in Management and Evaluation in Patients With Pleural Effusion
Status: Completed | Type: Observational
Sponsor: Deep Breeze (Industry)
Responsible Party: Merav Gat/VP Clinical Affairs, Deep Breeze
Other Study IDs: DB029
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; lung sounds; acoustic monitoring
MeSH Terms: conditions — Pleural Effusion; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with pleural effusion: Patients diagnosed with pleural effusion and presenting for treatment

SUMMARY:
The primary purpose of this study is evaluate the VRI device's accuracy in diagnosis of pleural effusion (in comparison to chest x-ray and ultrasonography), and to assess the pleural effusion location and size. The VRI system uses pressure sensors (electronic stethoscopes) to record the energy created by the airflow in the lungs during breathing.

DETAILED DESCRIPTION:
The accumulation of excess fluid in the pleural cavity of the lungs, known as pleural effusion, is a common clinical condition that may be the result of trauma or disease. Diagnosis and management of pleural effusion can be done by X-Ray or ultrasound; however X-Ray emits radiation, requires a special room and expert personnel, while ultrasound requires a high level of expertise to perform and analyze. The VRI device is non-invasive and radiation free. The VRI device is a simple method to image the lungs in a regional manner to examine changes that occur during pleural effusion.

Comparison: X-ray and ultrasonography evaluations of pleural effusion, compared to VRI acoustic imaging evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to read, understand, and provide written Informed Consent;
* Male or Female in the age range of 18-85 years;
* Subject is suspected to have pleural effusion;
* Body mass index (BMI) > 21.

Exclusion Criteria:

* Chest wall deformation;
* Spine deformation (including severe scoliosis);
* Hirsutism;
* Potentially contagious skin lesion on the back;
* Skin lesion that would interfere with sensor placement;
* Cardiac pacemaker or implantable defibrillator;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pleural effusion
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2006-11; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Ernst, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts, United States

REFERENCES:
- [Background] Marel M, Stastny B, Melinova L, Svandova E, Light RW. Diagnosis of pleural effusions. Experience with clinical studies, 1986 to 1990. Chest. 1995 Jun;107(6):1598-603. doi: 10.1378/chest.107.6.1598. PMID 7781353
- [Background] Heffner JE, Brown LK, Barbieri CA. Diagnostic value of tests that discriminate between exudative and transudative pleural effusions. Primary Study Investigators. Chest. 1997 Apr;111(4):970-80. doi: 10.1378/chest.111.4.970. PMID 9106577
- [Background] Mergo PJ, Helmberger T, Didovic J, Cernigliaro J, Ros PR, Staab EV. New formula for quantification of pleural effusions from computed tomography. J Thorac Imaging. 1999 Apr;14(2):122-5. doi: 10.1097/00005382-199904000-00011. PMID 10210486
- [Background] Dellinger RP, Jean S, Cinel I, Tay C, Rajanala S, Glickman YA, Parrillo JE. Regional distribution of acoustic-based lung vibration as a function of mechanical ventilation mode. Crit Care. 2007;11(1):R26. doi: 10.1186/cc5706. PMID 17316449